CLINICAL TRIAL: NCT04203797
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effect of Dupilumab on Exercise Capacity in Patients With Moderate-to-Severe Asthma
Brief Title: A Study to Evaluate the Effect of Dupilumab on Exercise Capacity in Adult Patients With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AS-1903; 2019-002742-20 (EudraCT Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dupilumab (Experimental): A loading dose at the start of the treatment followed by once every two weeks (Q2W).
  Interventions: Drug: dupilumab
- Matching placebo (Experimental): Matching dupilumab
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: dupilumab — Pre-filled syringe administered by subcutaneous (SC) injections
  Other Names: Dupixent®; SAR231893
  Arms: dupilumab
Drug: Matching placebo — Pre-filled syringe administered by subcutaneous (SC)
  Arms: Matching placebo

SUMMARY:
The primary objective of the study is to demonstrate that dupilumab treatment improves exercise capacity in patients with moderate-to-severe asthma.

The secondary objectives of the study are:

* To demonstrate that dupilumab treatment increases physical activity of daily living in patients with moderate-to-severe asthma
* To demonstrate that dupilumab treatment improves pre- and post-exercise lung function in patients with moderate-to-severe asthma

ELIGIBILITY:
Key Inclusion Criteria:

* A physician diagnosis of asthma
* Pre-bronchodilator FEV1 between 30% and 75% predicted at both the screening and baseline visits
* Bronchodilator reversibility defined as >200 mL and 12% increase in FEV1 post-administration of a short-acting beta agonist (SABA). A patient may also qualify if there is a documented history of bronchodilator reversibility or positive methacholine challenge test within 12 months prior to the screening visit
* Stable background therapy for at least 3 months with a stable dose ≥4 weeks prior to the baseline visit of a medium-to-high dose ICS (fluticasone propionate ≥250 to 1000 μg twice daily [BID] or equivalent) in combination with at least a second controller medication (eg, long-acting beta agonist [LABA], long-acting muscarinic antagonist [LAMA], leukotriene receptor antagonist [LTRA], theophylline, etc.); a third controller is allowed and with the same stabilization requirements
* Blood eosinophil count ≥300 cells/μL for patients not on maintenance OCS at the screening visit
* ACQ-5 score ≥1.5 at the screening and baseline visits

Key Exclusion Criteria:

* Body mass index >35 kg/m2 at screening
* Current smoking, vaping or tobacco chewing or cessation of any of these within 6 months prior to randomization, or >10 pack years smoking history
* Patients who require supplemental oxygen at screening
* Clinically significant cardiac disease as described in the protocol
* Uncontrolled hypertension at screening or baseline
* Participation in exercise or physical rehabilitation program within last 6 months prior to screening or planned during the study
* Previous use of dupilumab
* Anti-IgE therapy (eg, omalizumab [Xolair®]) within 130 days prior to visit 1 or any other biologic therapy (including anti-IL5, anti-IL-5R, anti-IL4Rα, anti-IL-13 mAb) or systemic immunosuppressant (eg, methotrexate, any anti-tumor necrosis factor mAbs, Janus kinase inhibitors, B- and/or T-cell targeted immunosuppressive therapies) to treat inflammatory disease or autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis) and other diseases, within 3 months or 5 half-lives prior to screening, whichever is longer
* Exposure to another investigative drug (monoclonal antibodies as well as small molecules) within a period prior to screening, of <3 months or <5 half-lives (whichever is longer)
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study
* Women of childbearing potential (WOCBP)* who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 12 weeks after the last dose

NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Management, Study Director — Regeneron Pharmaceuticals
Locations (30):
- United States (13):
  - Palos Verdes Medical Group (PVMG); Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - UCLA Medical Center - Harbor, Torrance, California
  - Allianz Research Institute, Westminster, California
  - University of Iowa Hospitals & Clinics-Roy J. and Lucille A. Carver College of Medicine, Iowa City, Iowa
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - American Health Research, Charlotte, North Carolina
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Regeneron Study Site, Hendersonville, Tennessee
  - The University of Texas Medical School at Houston, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
- France (3):
  - CHU Dijon, Dijon, Bourgogne-Franche-Comté
  - CHU Reims, Reims, Marne
  - CHU de Strasbourg - Nouvel Hopital Civil, Strasbourg
- Germany (9):
  - Praxis Dr. M. Rolke u. Dr. P. Rueckert, Aschaffenburg, Bavaria
  - Regeneron Study Site, Frankfurt am Main, Hesse
  - IKF Pneumologie GmbH & Co. KG - Institut fuer klinische Forschung Pneumologie Frankfurt (Clinical Research Centre Respiratory Medicine) to IKF Pneumologie Frankfurt GmbH & Co KG., Frankfurt am Main, Hesse
  - Regeneron Study Site, Hanover, Lower Saxony
  - Regeneron Study Site, Koblenz, Rhineland-Palatinate
  - IKF Pneumologie Mainz, Helix Medical Excellence Center Mainz, Mainz, Rhineland-Palatinate
  - Regeneron Study Site, Großhansdorf, Schleswig-Holstein
  - KLB - Gesundheitsforschung Luebeck GmbH, Lübeck, Schleswig-Holstein
  - Regeneron Study Site, Berlin
- Poland (3):
  - Regeneron Study Site, Lubin, Lower Silesian Voivodeship
  - Centrum Medycyny Oddechowej, Mroz Spolka Jawna, Bialystok
  - Lekarze Specjalisci - J. Malolepszy i Partnerzy, Wroclaw
- Spain (2):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Maranon (HGUGM) - Instituto de Investigacion Sanitaria Gregorio Maranon (IiSGM), Madrid

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (eg, FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 127 participants screened, 87 screen-fail, 40 participants randomized
Groups:
- Placebo: Matching dupilumab placebo
Period: Overall Study
Arm/Group | Placebo | Dupilumab
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Did not complete End of Study follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (7.7) | 45.3 (7.8) | 45.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Constant Work Rate Exercise Endurance Time - CWRET (Constant Work Rate Exercise Test)
Description: CWRET (Constant Work Rate Exercise Test) will be performed on an electromagnetically-braked cycle ergometer in an exercise physiology laboratory overseen by a trained pulmonologist or medical doctor designee.
Time Frame: Up to week 12
Population: The full analysis set (FAS) includes all randomized participants. The FAS is based on the treatment allocated (as randomized). Here 'n' = number of evaluable participants at a specified point in time.
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 17 | 20
Minutes | 0.923 [-0.614 to 2.460] | 1.742 [-0.054 to 3.538]

2. Secondary Outcome: Change From Baseline to Week 12 in Average Number of Steps Walked Per Day
Description: Based on accelerometry data
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 15 | 16
Steps | -1066.11 [-2921.32 to 789.10] | 925.92 [-691.46 to 2543.30]

3. Secondary Outcome: Change From Baseline to Week 12 in Total Energy Expenditure
Description: Metabolic equivalents of tasks [METs]. Based on accelerometry data
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: METs (metabolic equivalent of task)
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 15 | 16
METs (metabolic equivalent of task) | 23.40 [-87.37 to 134.17] | 59.36 [-15.83 to 134.55]

4. Secondary Outcome: Change From Baseline to Week 12 in the Mean Duration of Moderate-to-vigorous Physical Activity
Description: Defined as ≥3 METs. Based on accelerometry data
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 15 | 16
Minutes | -11.01 [-30.52 to 8.50] | 9.38 [-13.41 to 32.18]

5. Secondary Outcome: Change From Baseline to Week 12 in Pre- and Post-exercise Forced Expiratory Volume in One Second (FEV1)
Description: Based on spirometry data
Time Frame: Up to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 20 | 20
Liters
  Change from Baseline to Week 12 (Pre-exercise): number analyzed (Participants) | 16 | 20
  Change from Baseline to Week 12 (Pre-exercise) | 0.2123 [0.0072 to 0.4174] | 0.4205 [0.1409 to 0.7000]
  Change from Baseline to Week 12 (2-min Post-Exercise): number analyzed (Participants) | 3 | 4
  Change from Baseline to Week 12 (2-min Post-Exercise) | 0.2550 [-0.2390 to 0.7490] | 0.2902 [0.0886 to 0.4919]
  Change from Baseline to Week 12 (5-min Post-Exercise): number analyzed (Participants) | 14 | 17
  Change from Baseline to Week 12 (5-min Post-Exercise) | 0.2416 [0.0238 to 0.4593] | 0.4156 [0.1505 to 0.6808]
  Change from Baseline to Week 12 (10-min Post-Exercise): number analyzed (Participants) | 15 | 18
  Change from Baseline to Week 12 (10-min Post-Exercise) | 0.2211 [0.0180 to 0.4243] | 0.4613 [0.2167 to 0.7060]
  Change from Baseline to Week 12 (20-min Post-Exercise): number analyzed (Participants) | 15 | 20
  Change from Baseline to Week 12 (20-min Post-Exercise) | 0.2496 [0.0608 to 0.4384] | 0.4738 [0.2230 to 0.7245]

ADVERSE EVENTS:
Time Frame: Up to 22 weeks
Groups:
- Dupilumab 300 mg Q2W: A loading dose at the start of the treatment followed by once every two weeks (Q2W).
Arm/Group | Placebo | Dupilumab 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Dupilumab 300 mg Q2W (N=20)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT04203797/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04203797/SAP_001.pdf